CLINICAL TRIAL: NCT04520113
Title: Innovative Contact Tracing Strategies for Detecting TB in Mobile Rural and Urban South African Populations
Brief Title: Kharituwe TB Contact Tracing Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Perinatal HIV Research Unit of the University of the Witswatersrand (Other); Setshaba Research Centre (Unknown); The National Institute for Communicable Diseases (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: R01AI147681 (NIH); IRB00011124 (Other: JHSPH IRB)
Record Dates: First submitted 2020-08-07; First posted 2020-08-20 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Tuberculosis; Hiv
MeSH Terms: conditions — Tuberculosis; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The principal investigators are blinded as to the assignment of treatment to participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Tracing (Active Comparator): Households of tuberculosis index patients receive "standard" household contact tracing during regular weekday business hours.
  Interventions: Behavioral: Household contact tracing
- Holiday Tracing (Experimental): Households of tuberculosis index patients in rural South Africa receive household contact tracing during holidays (Christmas and Easter).
  Interventions: Behavioral: Household contact tracing
- Evening / Weekend Tracing (Experimental): Households of tuberculosis index patients in urban South Africa receive household contact tracing during evenings and weekends.
  Interventions: Behavioral: Household contact tracing

INTERVENTIONS:
Behavioral: Household contact tracing — Household contact tracing to test and diagnose Tuberculosis of household contacts of Tuberculosis patients.

SUMMARY:
The purpose of this study is to characterize the role of human mobility in fueling TB epidemics and estimate the potential impact of innovative case finding interventions tailored to mobile populations

DETAILED DESCRIPTION:
The investigators propose a randomized trial of two novel TB case-finding interventions among household members of patients diagnosed with active TB: holiday-based screening in a rural South African province (Limpopo) and off-peak (weekend/evening) screening in an urban settlement into which many residents of Limpopo migrate for work. The investigators will enroll index cases of TB plus their household contacts in each setting and randomize them to novel versus standard contact investigation. In Specific Aim 1, investigators will use whole genome sequencing of all cases, overlaying transmission trees with data on human movement, to evaluate associations between mobility and TB transmission in this population. In Specific Aim 2, investigators will employ a multidisciplinary approach to compare novel versus standard contact investigation in each setting along the following dimensions: (a) effectiveness (number of secondary TB cases diagnosed and starting treatment); (b) implementation (reach, fidelity, and maintenance of contact investigation outside of business hours); (c) cost-effectiveness (cost per disability-adjusted life year) and budget impact; and (d) projected population-level impact on TB incidence. Successful completion of these aims will have long-term impact by characterizing the role of mobility in fueling TB epidemics and testing two tailored approaches to improve TB control in highly mobile populations - an underserved group that is increasingly recognized as playing a major role in global TB transmission.

ELIGIBILITY:
TB index cases:

Inclusion criteria:

* Age 0-99 years (Including those recently deceased)
* Diagnosed with pulmonary TB at a study hospital or clinic (microbiological and/or chest x-ray diagnosis)

Exclusion criteria:

* Unwilling/unable to provide informed consent (including next of kin, for those recently deceased)
* Plan not to pursue TB treatment within the study district
* Unwilling/unable to comply with study procedures

Contacts:

Inclusion criteria:

* Age 0-99 years
* Currently resides with or visiting eligible TB index case

Exclusion Criteria:

* Unwilling/unable to provide informed consent
* Unwilling/unable to comply with study procedures

Max Age: 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10579 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W. Dowdy, MD, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- South Africa (2):
  - Perinatal HIV Research Unit (PHRU), Johannesburg
  - Setshaba Research Centre, Soshanguve

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hanrahan CF, Nonyane BAS, Biche P, Mohlamonyane M, Morolo M, Omar SV, Ahmed K, Martinson N, Dowdy DW. Timing of household contact investigation for tuberculosis among rural and urban populations in South Africa (Kharituwe study): a pragmatic individually randomized controlled trial. EClinicalMedicine. 2026 Jan 16;91:103744. doi: 10.1016/j.eclinm.2025.103744. eCollection 2026 Jan. PMID 41607590
- [Derived] Young N, Biche P, Mohlamonyane M, Morolo M, Maholwana B, Ahmed K, Martinson N, Hanrahan CF, Dowdy DW. Innovative timing strategies for tuberculosis household contact investigation: cost-effectiveness analysis from a randomized trial in rural and urban South Africa (Kharituwe Study). EClinicalMedicine. 2025 May 26;84:103259. doi: 10.1016/j.eclinm.2025.103259. eCollection 2025 Jun. PMID 40503514
- [Derived] Mlambo LM, Milovanovic M, Hanrahan CF, Motsomi KW, Morolo MT, Mohlamonyane MP, Albaugh NW, Ahmed K, Martinson NA, Dowdy DW, West NS. The impact of ethical implications intertwined with tuberculosis household contact investigation: a qualitative study. medRxiv [Preprint]. 2024 Jun 28:2024.06.27.24309538. doi: 10.1101/2024.06.27.24309538. PMID 38978659

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive eligible index participants with TB were recruited from among 12 public hospitals in Limpopo and 33 primary health care clinics and 2 public hospitals in Soshanguve.
Pre-assignment Details: The actual enrollment in the study contains the 4417 index TB cases, and within the index participants' households, 6162 contact persons, for a total of 10579 enrolled individuals. Only the 4417 index TB cases were randomized to arms.
Groups:
- Standard Tracing- Limpopo: This arm was located in the Limpopo site. Households of tuberculosis index patients receive "standard" household contact tracing during regular weekday business hours.
  Household contact tracing: Household contact tracing to test and diagnose Tuberculosis of household contacts of Tuberculosis patients.
- Standard Tracing- Soshanguve: This arm was located in the Soshanguve site. Households of tuberculosis index patients receive "standard" household contact tracing during regular weekday business hours.
  Household contact tracing: Household contact tracing to test and diagnose Tuberculosis of household contacts of Tuberculosis patients.
Period: Overall Study
Arm/Group | Standard Tracing- Limpopo | Holiday Tracing | Evening / Weekend Tracing | Standard Tracing- Soshanguve
Started | 4368 | 1952 | 1320 | 2939
TB Index Cases | 1335 | 666 | 804 | 1612
Contact Persons | 3033 | 1286 | 516 | 1327
Completed | 4368 | 1952 | 1320 | 2939
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Index TB and contact person participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Tracing- Limpopo | Holiday Tracing | Evening / Weekend Tracing | Standard Tracing- Soshanguve | Total
Number analyzed (Participants) | 4368 | 1952 | 1320 | 2939 | 10579
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: The rows detail the two populations who make up the overall population-- TB index participants and Contact person participants
  years
    Index TB participants: number analyzed (Participants) | 1335 | 666 | 804 | 1612 | 4417
    Index TB participants | 41 [31 to 51] | 42 [32 to 53] | 42 [30 to 52] | 41 [31 to 53] | 41 [31 to 52]
    Contact person participants: number analyzed (Participants) | 3033 | 1286 | 516 | 1327 | 6162
    Contact person participants | 18 [6 to 37] | 18 [6 to 40] | 33 [19 to 55] | 34 [21 to 55] | 27 [9 to 43]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The rows detail the two populations who make up the overall population-- TB index participants and Contact person participants
  Participants
    Index TB participants: number analyzed (Participants) | 1335 | 666 | 804 | 1612 | 4417
    Index TB participants: Female | 584 | 286 | 330 | 566 | 1766
    Index TB participants: Male | 751 | 380 | 474 | 1046 | 2651
    Contact person participants: number analyzed (Participants) | 3033 | 1286 | 516 | 1327 | 6162
    Contact person participants: Female | 1884 | 785 | 346 | 849 | 3864
    Contact person participants: Male | 1149 | 501 | 170 | 478 | 2298
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The rows detail the two populations who make up the overall population-- TB index participants and Contact person participants
  Participants
    Index TB Participants: number analyzed (Participants) | 1335 | 666 | 804 | 1612 | 4417
    Index TB Participants: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Index TB Participants: Asian | 0 | 0 | 0 | 0 | 0
    Index TB Participants: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Index TB Participants: Black or African American | 1325 | 666 | 801 | 1601 | 4393
    Index TB Participants: White | 0 | 0 | 0 | 0 | 0
    Index TB Participants: More than one race | 10 | 0 | 3 | 11 | 24
    Index TB Participants: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
    Contact person participants: number analyzed (Participants) | 3033 | 1286 | 516 | 1327 | 6162
    Contact person participants: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Contact person participants: Asian | 0 | 0 | 0 | 0 | 0
    Contact person participants: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Contact person participants: Black or African American | 3020 | 1285 | 514 | 1325 | 6144
    Contact person participants: White | 0 | 0 | 0 | 0 | 0
    Contact person participants: More than one race | 13 | 1 | 2 | 2 | 18
    Contact person participants: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa: Index TB Participants | 1335 | 666 | 804 | 1612 | 4417
  South Africa: Contact person participants | 3033 | 1286 | 516 | 1327 | 6162

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness: Mean Number of Secondary TB Cases Identified and Started on Treatment Per Index Case in Each Arm
Description: The mean number of secondary TB cases identified and started on treatment per index case for each arm.
Time Frame: Up to 35 months
Measure: Mean (95% Confidence Interval); unit: mean secondary TB cases
Groups:
- Holiday Tracing: This arm was located in the Limpopo site. Households of tuberculosis index patients in rural South Africa receive household contact tracing during holidays (Christmas and Easter).
  Household contact tracing: Household contact tracing to test and diagnose Tuberculosis of household contacts of Tuberculosis patients.
- Evening / Weekend Tracing: This arm was located in the Soshanguve site. Households of tuberculosis index patients in urban South Africa receive household contact tracing during evenings and weekends.
  Household contact tracing: Household contact tracing to test and diagnose Tuberculosis of household contacts of Tuberculosis patients.
Arm/Group | Standard Tracing- Limpopo | Holiday Tracing | Evening / Weekend Tracing | Standard Tracing- Soshanguve
Number analyzed (Participants) | 4368 | 1952 | 1320 | 2939
mean secondary TB cases | 1.7 [0.9 to 2.5] | 1.2 [0.5 to 1.9] | 2.3 [1.0 to 3.2] | 2.4 [1.8 to 3.0]

2. Secondary Outcome: The TB Prevalence Ratio, Comparing Highly Mobile to Less Mobile Index Patients
Description: The TB prevalence ratio, comparing highly mobile to less mobile individuals, measuring mobility on two scales (neighborhood/intra-urban and regional/intra-national). For the analysis: amount of time spent in transit, truncating long excursions at 50km (one hour).
Time Frame: Duration of study (30 months)
Reporting Status: Not Posted

3. Secondary Outcome: TB Strain Relatedness Using Maximum Likelihood Transmission Trees.
Description: TB natural history, epidemiological, and whole genome sequencing (WGS)-derived phylogenetic data will be integrated into a statistical modeling framework to draw probabilistic conclusions about the likelihood of transmission between persons. "Transmitters" will be defined as individuals from whom at least one secondary case most likely originated.
Time Frame: Duration of study (30 months)
Reporting Status: Not Posted

4. Secondary Outcome: Relative Acceptability of Each Novel Strategy Compared to Standard Contact Investigation
Description: Relative acceptability of each novel strategy, compared against routine contact investigation. Acceptability of the intervention will be measured among index cases and contacts using a short questionnaire given to a randomly selected participant at a randomly selected 15% of the households visited. The interview will cover acceptability of the visit timing, notification, visit activities (TB screening, HIV testing) and study team interaction among others.
Time Frame: Duration of study (30 months)
Reporting Status: Not Posted

5. Secondary Outcome: Feasibility of Each Strategy: Proportion of Potentially Eligible Index Cases for Whom a Household Visit Was Conducted
Description: Feasibility of each strategy as the proportion of potentially eligible index cases for whom a household visit was conducted. All reasons why visits were unable to be conducted will be recorded (e.g. could not find household, no one ever home, visit not conducted during expected off-peak period).
Time Frame: Duration of study (30 months(
Reporting Status: Not Posted

6. Secondary Outcome: Relative Fidelity of Each Novel Strategy Compared to Standard Contact Investigation
Description: Relative fidelity of each novel strategy using a process checklist for each index case and household, including whether the household visit was offered and accepted, whether the visit was attempted, whether the visit was successful (i.e., enrolled at least one contact), whether symptom screening and sputum collection were completed and whether newly identified TB cases were notified and referred for treatment.
Time Frame: Duration of study (30 months)
Reporting Status: Not Posted

7. Secondary Outcome: Sustainability of Each Novel Strategy Relative to Standard Contact Tracing
Description: Sustainability of each novel strategy by reporting the primary outcome and fidelity measures according to six-month time period over the course of the study.
Time Frame: Duration of study (30 months)
Reporting Status: Not Posted

8. Secondary Outcome: Incremental Cost-effectiveness Ratio for Each Novel Strategy Relative to Standard Contact Tracing
Description: Defined as (cost of contact tracing strategy 2 - cost of strategy 1)/(effectiveness of strategy 2 - effectiveness of strategy 1), where effectiveness is modeled as the number of disability-adjusted life years (DALYs) averted by the intervention. The primary cost-effectiveness measures will be the incremental cost per DALY averted using novel strategies (holiday and off-hours contact tracing) compared to routine contact tracing in each setting separately.
Time Frame: Duration of study (30 months)
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Adverse Events were not collected
Arm/Group | Standard Tracing- Limpopo | Holiday Tracing | Evening / Weekend Tracing | Standard Tracing- Soshanguve
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT04520113/Prot_SAP_001.pdf